CLINICAL TRIAL: NCT02715427
Title: Enhanced Recovery After Hepatic Surgery Versus Conventional Care : a Controlled Randomized Monocentric Trial (MultiPAS).
Brief Title: Enhanced Recovery After Hepatic Surgery (MultiPAS).
Acronym: MultiPAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-A01806-43
Record Dates: First submitted 2016-03-11; First posted 2016-03-22 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-04

CONDITIONS: Liver Surgery
MeSH Terms: interventions — Enhanced Recovery After Surgery

ARMS (2):
- Conventional care (Active Comparator): Preoperative consultation Information support conventional perioperative No bowel preparation
  Day before surgery Normal diet until midnight No carbohydrate loading Premedication with anxiolytic
  Operative day Conventional general anaesthesia Classic management perfused volumes Conventional use of drains at the operative site Standard nasogastric drainage Conventional analgesia protocol
  Postoperative time Mobilization from J1 Progressive refeeding Progressive removal of venous, arterial and urinary catheters. Gradual recovery of the usual treatment from J1 Breathe physiotherapy depending on the clinical course No stimulation of intestinal transit
  Interventions: Other: Conventional care
- Enhanced recovery (Experimental): Preoperative consultation Specific information about the enhanced rehabilitation No bowel preparation Immunonutrition for the 7 preoperative days
  Day before surgery Minimal preoperative fasting No premedication Carbohydrate loading
  Operative day Optimized general anesthesia Reduced volumes perfused Limiting use of drains at the operative site Reduced doses of morphine Local anesthetic usage No standard use of nasogastric drainage
  Postoperative time Stimulation mobilization from D0 Refeeding "on demand " from D0 Early removal of venous, arterial and urinary catheters. J1 recovery from the majority of the usual treatment Breathe physiotherapy from D0 to D5 Ileus prevention by chewing gum
  Interventions: Other: Enhanced recovery

INTERVENTIONS:
Other: Conventional care
  Arms: Conventional care
Other: Enhanced recovery
  Arms: Enhanced recovery

SUMMARY:
Enhanced rehabilitation programs are based on new therapies and treatment combinations to reduce the length of hospitalization, duration of postoperative convalescence, morbidity, but also the overall cost of care. The operating stress and hypercatabolic conditions surrounding the surgery are sources of complications. In this enhanced rehabilitation approach, the principle is to fight through a series of actions against this surgical stress. Several North American studies, Chinese, Scandinavian or Batavian have shown the feasibility and the interest of enhanced perioperative rehabilitation in liver surgery. Nevertheless, there is not until now French data concerning the assessment of enhanced rehabilitation in liver surgery. The main objective of the study is to compare the effectiveness of the implementation of a multimodal management program after liver surgery in a French university center compared to conventional care. Secondary objectives of the study are to compare an enhanced rehabilitation program in liver surgery versus conventional treatment in terms of morbidity and mortality in the immediate postoperative period and until day 90, length of hospital stay, blood loss and the delay to bowel mobility recovery. Compliance to the program in both groups will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patient to be operated on for hepatectomy in Universitary Hospital of Angers
* No emergency surgery
* No bilio-digestive anastomosis
* Body Mass Index between 18 and 40 kg/m2
* Preoperative morbidity status graded with the American Society of Anesthesiologists (ASA) between I to III
* Affiliated to the national health insurance

Exclusion Criteria:

* Pregnant woman
* Patient who doesn't speack french
* Colorectal surgery combined
* Postoperative stay predictable in critical care unit
* Patient under law protection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Day number to functional recovery | 90 days
  The evaluation of time to functional recovery is scored once a day. A patient is fully functionally recovered when all of the following criteria are satisfied:
  1. adequate pain control with oral analgesia: Post-operative pain is rated by the numeric rating scale. Nurses ask patients the intensity of their current pain on a scale of 0 (no pain) to 10 (worst possible pain). To satisfy this criterion, patient must rate their pain between 0 to 3 with only oral analgesics.
  2. restoration of mobility to an independent level We decided to use the Groningen Activity Restriction Scale for rated the difference between preoperative and postoperative mobility level. To satisfy this criterion, patient must have the same score in postoperative.
  3. absence of intravenous fluid administration for at least 24 hours.
  4. ability to eat solid foods well tolerated for at least 24 hours to satisfy this criterion.
  5. normal or decreasing serum bilirubin level and international normalised ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, Maine et Loire, France